CLINICAL TRIAL: NCT06116656
Title: Changes in Host Gene Expression to Differentiate Between Systemic Inflammation and Infection After Major Surgery
Acronym: PAX
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: Amphia Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, associate professor, St. Antonius Hospital
Other Study IDs: NL
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Infections; Sepsis
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected in PAX gene blood RNA tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood leucocyte transcriptomics — the analysis of the RNA transcripts produced by the genotype at a given time that provides a link between the genome, the proteome, and the cellular phenotype.
  Other Names: not apllicable

SUMMARY:
Changes in host gene expression may provide additional information to diagnose postoperative infection and improve outcome after surgery. This study aims to validate the early diagnostic performance of specific gene signatures for differentiating infection from non-infected SIRS or uncomplicated postoperative course in blood sampes of adult patients undergoing major noncardiac surgery.

DETAILED DESCRIPTION:
Rationale: Differentiation between the systemic inflammatory response syndrome (SIRS) and infection after surgery is challenging. Consequent diagnostic uncertainty may result in delayed diagnosis and interventions to prevent organ dysfunction or eventually death. Changes in host gene expression may provide additional information to diagnose postoperative infection and improve outcome after surgery.

Objective: To validate the early diagnostic performance of specific gene signatures1 for differentiating infection from non-infected SIRS or uncomplicated postoperative course.

Study design: A prospective observational multicenter study. Study population: Adult patients undergoing major noncardiac surgery. Main study parameters/endpoints: Main study parameters are specific gene signatures. Main study endpoint is postoperative infection and SIRS.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In each patient blood samples will be drawn for analysis on the following time points: after induction for anaesthesia, directly postoperative and on postoperative day 1 - 7. For each sample 2.5 ml of blood is taken. In a total of 9 samples this results in a cumulative volume of 22.5 ml. Whenever possible, blood samples will be drawn simultaneously with routine perioperative laboratory testing. In case of admission to the Intensive Care Unit blood samples will be collected using an arterial line. There are no direct risks or benefits for patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Major noncardiac surgery with infection risk >20%

Exclusion Criteria:

* Age <18 years
* Emergency surgery
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major noncardiac surgery with infection risk >20%
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative infection | 30 days
  Infection after surgery

SECONDARY OUTCOMES:
Postoperative SIRS | 30 days
  SIRS after surgery
Postoperative sepsis | 30 days
  Sepsis after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia hospital, Breda
  - St Antonius hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No